#### Goal

The aim of this study is to evaluate the effect of breastfeeding education given by teach-back method on breastfeeding success.

# **Hypotheses**

H0: Breastfeeding training given by Teach-Back method has no effect on breastfeeding success.

H1: Breastfeeding training given by Teach-Back method has an impact on breastfeeding success.

### Methods

# Study design

This study, which has a randomized controlled experimental research design, was conducted between 15 January and 15 December 2018. The sample of the study was divided into two groups by randomization. Breastfeeding success levels were compared by providing breastfeeding education and counseling service based on the teach-back method to one group of mothers (intervention group), and standard breastfeeding education and counseling service to another group (control group). Opinions were received from five academicians working in the field of Midwifery, Obstetrics and Gynecology Nursing, who have researches on breastfeeding. Recommendations from the CONSORT group (Consolidated Standards of Reporting Trials) were followed in this study (Schulz et al., 2010).

# Sample and setting

Women who lives in a city center where is in Turkey's Central Anatolia and have a vaginal birth, literate, primipar, in term and healthy. Those excluded from the inclusion criteria were excluded from the study.

The study was carried out in the City Hospital, where the number of births in the city center was the highest in a year, and in the Family Health Centers where maternal and infant follow-ups were performed. The first stage of the study, which was the stage of meeting women, was done in the maternity unit and postpartum service of the City Hospital, since women who gave vaginal births were

discharged after 24 hours if no problem developed. The second stage of the study was carried out in Family Health Centers where women are affiliated.

# Sample size calculation

The universe of the study was composed of women who had vaginal births in the City Hospital between years 2017-2018. According to the hospital records, in the first 6 months of 2017, the total number of births was determined as 1455, and the number of non-invasive vaginal births was 590. The minimum number of individuals to be included in the sample of the study was calculated using the "G-power 3.1.3" program based on the data of the study titled "The effect of antenatal training based on strengthening breastfeeding self-efficacy perception and breastfeeding success" (Tokat Aluş & Okuş , 2013). Considering the sample size of the research and the mean scores obtained from this study, the LACTH scale scores will increase 0.5 points after the application, with the pre-acceptance of the clinical effect to be 5% of Alpha error and 80% of the power of the study (Effect Size: 0.70) and it was determined that there should be at least 31 people in each group (Tokat Aluş & Okumuş, 2013). A total of 80 women, 40 studies and 40 control groups, were included in the sample. Women who had vaginal births meeting the inclusion criteria were selected by simple random randomization into the intervention and control group.

# Randomization

Considering the inclusion and exclusion criteria, women were divided into simple randomization intervention and control groups. In the randomization of the sample, "Research Randomizer" was used. The randomization process was created by a neutral researcher who was not involved in the study. The women were not informed about the groups they were in. Single blind was provided in the study by knowing which group they would be in by the researcher.

### Intervention

The study was carried out in two stages. In the first stage, in the first 24 hours at the postpartum period, the researcher interviewed the women who gave birth in the postpartum care units of the hospital and

determined the women who volunteered to participate in the research and that comply with the inclusion criteria and received their informed consent. Women were divided into randomized intervention or control groups. When the postpartum mother and baby's health condition was stable, "Personal Information Form" was applied to mothers. After the women were informed about the appointments and dates at the Family Health Centers where the second phase of the research will be carried out, the home and mobile numbers of the researcher were given to them in writing. The meeting ended with the mothers about the time and place of the next visits.

In the second stage of the study, three interviews were held with the mothers on the dates determined in the first stage of the study. In these interviews, the mothers in the intervention group were asked by the researchers about the needs of breastfeeding by using the relevant literature (Ekşioğlu, 2016; Hannula, Kaunonen, & Tarkka, 2008; Maleki-Saghooni et al., 2017; RNAO, 2018). Training and counseling based on the Teach-back method was given in the Family Health Centers (FHC) where they are registered. Turkey Ministry of Health's Postpartum Care Management Guidelines (2014) was carried out with mothers enrolled in FHC in the control group, on the basis of three interviews. In these interviews, standard training and counseling services were offered on breastfeeding. While providing standard training and counseling services, "Breastfeeding Training Guide" used in the intervention group was taken as the basis. The method of straight expression, which is mostly used by breastfeeding counseling provider healthcare professionals in Turkey, was used. In standard education, whether the learning is achieved is tested by closed-ended, "yes-no" questions structured as "Did you understand?". After, it is controlled by asking whether there are any questions about the subject. The trainings of both groups were given individually in a separate room at FHCs.

#### Measurements and data collection

Based on the literature information (Faridvand, Mirghafourvand, Malakouti, & Mohammad-Alizadeh-Charandabi, 2017; Jeon & Hwang, 2013; Maleki-Saghooni et al., 2017; Tarrant, Younger, Sheridan-Pereira, & Kearney, 2011) an information form was developed by researchers. The form consisted of a total of 28 questions, including the socio-demographic and personal characteristics of women in the intervention and control group (16 questions), questions related to birth, postpartum period and

breastfeeding (12 questions). "LATCH Breastfeeding Diagnosis and Evaluation Scale" and "Postpartum Breastfeeding Self-Efficacy Scale Short Form" were used to evaluate breastfeeding success. The Breastfeeding Training Guide used in the education of mothers was created by scanning the literature on the subject (Aittasalo et al., 2006; Badaczewski et al., 2017; Farris, 2015; Tamura-Lis, 2013; Tokat, Okumuş, & Dennis, 2010) and in line with the recommendations of 5 academics specialized in Obstetrics and Gynecology Nursing. In order to evaluate the performance of the researcher using the Teach-back method, the "Teach-Back Method Observation Tool" recommended by the developers of this method was used.

# **Data Collection**

In the first stage of the study, women were interviewed in postpartum care units, and when the health condition of the mother and baby was stable, the Personal Information Form was applied to the mothers.

In the second stage of the study, 3 interviews were conducted with the mothers in the intervention and control groups during the 2-5th postpartum days, 13-17th days and 30-42nd days. In the first meeting of the second phase, the pre-education Breastfeeding Diagnostic Tool LATCH and Postpartum Breastfeeding Self-Efficacy Scale were applied to the mothers in the intervention and control groups. Breastfeeding training and counseling services were provided to the mothers in the intervention group, based on the teach-back method, and those in the control group using the standard breastfeeding training technique. This interview lasted an average of 1 hour.

In the second meeting of the second stage, which was held between the 13th and 17th days of birth, the pre-education Breastfeeding Diagnostic Tool LATCH and Postpartum Breastfeeding Self-Efficacy Scale were applied to the mothers in the intervention and control groups. Breastfeeding training and counseling services were provided to the mothers in the intervention group, based on the teach-back method, and those in the control group using the standard breastfeeding training technique. This interview took an average of 40-45 minutes.

In the third meeting of the second stage, which was held between the 30-42th days of birth, the preeducation Breastfeeding Diagnostic Tool LATCH and Postpartum Breastfeeding Self-Efficacy Scale were applied to the mothers in the intervention and control groups. Breastfeeding training and counseling services were provided to the mothers in the intervention group, based on the teach-back method, and those in the control group using the standard breastfeeding training technique. This interview took an average of 40-45 minutes.

### Statistical analysis

The data of the study were evaluated on computer by using Statistical Package for Social Sciences (SPSS) (22.0) program. In the evaluation of the data;

- The distribution of the data was evaluated with the Kolmogorov-Smirnov test. Since it showed a normal distribution, parametric tests were used in the analyzes.
- The homogeneity of the groups was assessed by chi-square test in categorical variables, Mann Whitney U in numerical variables, or T test in independent groups.
- In the intervention and control groups, "Multifaceted Variance Analysis in Repeated Measurements" was performed in comparing the LATCH breastfeeding diagnosis and evaluation scale and the breastfeeding self-efficacy scale according to the group, time and group \* time interaction.
- In the advanced analysis of the difference between the LATCH, breastfeeding diagnostic and evaluation scale, and breastfeeding self-efficacy scale averages in the intervention and control groups, "One-Way Variance Analysis in Repetitive Measurements" to compare the mean scores of the groups within themselves, "Bonferroni Correction Dependent Groups T-Test" to compare the measurements with each other.

# **Ethical consideration**

Before starting the research, permission was obtained from the Konya Chamber of Commerce, Karatay University Rectorate Medical Faculty Non-Device Research Ethics Committee (Date: 26.12.2017 and Number no: 006). Institution permissions were obtained from Yozgat City Hospital (Date: 05.02.2018 and Number: 78.535.428-799) and Provincial Health Directorate Family Health Unit (Date: 11.06.2018 and Number: 92.198.657-060.11.01).